CLINICAL TRIAL: NCT06566898
Title: Monitoring of Antimicrobial Resistance Based on Metagenomics Analyses in Pneumonia Patients: a Genomic Epidemiology Study
Brief Title: Monitoring of Antimicrobial Resistance Based on Metagenomics Analyses in Pneumonia Patients
Status: Recruiting | Type: Observational
Sponsor: Shanghai General Hospital, China (Other)
Collaborators: Wuxi People's Hospital Affiliated to Nanjing Medical University (Unknown); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); The Central Hospital of Huanggang (Other)
Responsible Party: Principal Investigator, Mei Kang, Principal Investigator, Shanghai General Hospital, China
Other Study IDs: 2023234
Record Dates: First submitted 2024-08-18; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Pneumonia; Next-generation Sequencing; Microbiome; Antimicrobial Resistance
Keywords: Pneumonia; Next-generation sequencing; Microbiome; Antimicrobial Resistance
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Nasopharyngeal swab, oropharyngeal swab, bronchoalveolar lavage fluid, sputum, blood, hydrothorax, lung tissue.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Severe pneumonia: Patients clinically diagnosed as severe pneumonia are diagnosed according to the Guidelines for the diagnosis and Treatment of community-acquired pneumonia in Adults (2019 edition) formulated by the American Thoracic Society (ATS) and the Infectious Diseases Society of America (IDSA), who meet 1 of the following major criteria or ≥3 minor criteria can be diagnosed. The diagnostic criteria for severe pneumonia in children were adopted by the British Thoracic Society (BTS) in 2011.
- Mild pneumonia: Patients clinically diagnosed as severe pneumonia and mild pneumonia are diagnosed according to the Guidelines for the diagnosis and Treatment of community-acquired pneumonia in Adults (2019 edition) formulated by the American Thoracic Society (ATS) and the Infectious Diseases Society of America (IDSA). The diagnostic criteria for severe and mild pneumonia in children were adopted by the British Thoracic Society (BTS) in 2011

SUMMARY:
Monitoring of antimicrobial resistance (AMR) based on metagenomics analyses in pneumonia patients is critical for optimizing clinical diagnosis and treatment and improving clinical prognosis. This study is designed to ask the following key questions:

1. What is the microbiome maps of patients with severe pneumonia and mild pneumonia ?
2. How many pathogen resistance genes are carrying in severe pneumonia and mild pneumonia ?
3. What is the genetic diversity of key pathogens detected in severe pneumonia and mild pneumonia during 2019-2025?

DETAILED DESCRIPTION:
This is a historical prospective obsevational study. Patients diagnosed with severe and mild pneumonia are recruited continously from four hospitals (Shanghai General Hospital, Wuxi People's Hospital Affiliated to Nanjing Medical University, Wuhan Union Hospital, and Huanggang Central Hospital) in China during March, 2019 to March, 2025.

Next-generation sequencing: Metagenomics and metatranscriptomic libraries undergo next-generation sequencing using the Illumina Novaseq 6000 platform.

Microbiome analysis: using KneadData (v0.10.0) reference from the human genome (GRCH38 reference database) to filter out the quality control of illumina sequencing data in Virosaurus download virus genome data sets for reference, bowtie2 (v2.3.4.1) (genome coverage >30%, depth >1X) was used to locate and analyze the post-host sequence, and then the "samtools idxstats" command was used to calculate the classification and relative abundance of viruses. Meanwhile, in order to obtain the annotation information of bacteria at the species level, PhyloFlash (v3.4) was used to calculate read counts for 16S rRNA genes in the SILVA database, selecting similarity greater than or equal to 98% as a threshold. Using eukaryotic pathogen genome database EUPATHDB46 as reference, bowtie2 and samtools were used for qualitative and quantitative analysis of fungal pathogens.

The criteria for determining the cause of respiratory infection are: (1) existing species known to be associated with human disease (ICD-10), (2) previously unidentified potential novel pathogens (only DNA and RNA viruses whose genera or families have previously been shown to infect mammals), and (3) possible symbiotic bacteria not included.

Analysis of AMR: by comparing the sequence similarity between the sequencing fragments and known drug resistance genes, the detection content can determine whether drug resistance genes exist, and suggest drug resistance caused by modification, inactivation, repression and other drug resistance genes.

Drug resistance genes detection: genes related to drug resistance recorded in CARD (Comprehensive Antibiotic Resistance Database) and ARG-ANNOT database. In this assay, only functional genes with drug resistance activities such as modification, inactivation, and repression, as well as pathway and target changes caused by some point mutations, were reported.

Genetic diversity was computed as the mean pairwise genetic distance within a group. Maximum likelihood phylogenetic trees were constructed using RaxML with a general time-reversible nucleotide substitution model and 1000 bootstraps. The genetic distance between sequences was calculated using MEGAX, with a bootstrap method for variance estimation.

ELIGIBILITY:
Inclusion Criteria:

* Patients clinically diagnosed as severe pneumonia and mild pneumonia are diagnosed according to the Guidelines for the diagnosis and Treatment of community-acquired pneumonia in Adults (2019 edition) formulated by the American Thoracic Society (ATS) and the Infectious Diseases Society of America (IDSA), who meet 1 of the following major criteria or ≥3 minor criteria can be diagnosed. The diagnostic criteria for severe and mild pneumonia in children were adopted by the British Thoracic Society (BTS) in 2011.
* Clinical examination was performed, and there was biospecimen (nasopharyngeal swab, oropharyngeal swab, bronchoalveolar lavage fluid, sputum, blood, hydrothorax, lung tissue) remaining in the clinical microbiological examination.

Exclusion Criteria:

* Patients whose biological samples may be contaminated;
* Patients with alveolar lavage fluid or hydrothorax volume less than 200μl.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pneumonia patients from four centers in China during 2022-2025.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Microbiome composition | during the study period, 2019-2025
  a collection of microbial communities detected in the biospecimen

SECONDARY OUTCOMES:
Alpha diversity | during the study period, 2019-2025
  the diversity within a particular area or ecosystem
Prevalence of bacterial resistance genes | during the study period, 2019-2025
  the number of bacterial resistance genes divided by the number of biospecimen
Beta diversity | during the study period, 2019-2025
  a comparison of of diversity between ecosystems, usually measured as the amount of species change between the ecosystems

CONTACTS AND LOCATIONS:
Overall Officials: Mei Kang, MPH, Principal Investigator — Shanghai General Hospital, Shanghai Jiaotong University School of Medicine
Locations (1):
- Mei Kang, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
The datasets used in this study are available upon request to the principle investigator.

REFERENCES:
- [Background] GBD 2019 Diseases and Injuries Collaborators. Global burden of 369 diseases and injuries in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2020 Oct 17;396(10258):1204-1222. doi: 10.1016/S0140-6736(20)30925-9. PMID 33069326
- [Background] File TM Jr, Ramirez JA. Community-Acquired Pneumonia. N Engl J Med. 2023 Aug 17;389(7):632-641. doi: 10.1056/NEJMcp2303286. No abstract available. PMID 37585629
- [Background] Limmathurotsakul D, Dunachie S, Fukuda K, Feasey NA, Okeke IN, Holmes AH, Moore CE, Dolecek C, van Doorn HR, Shetty N, Lopez AD, Peacock SJ; Surveillance and Epidemiology of Drug Resistant Infections Consortium (SEDRIC). Improving the estimation of the global burden of antimicrobial resistant infections. Lancet Infect Dis. 2019 Nov;19(11):e392-e398. doi: 10.1016/S1473-3099(19)30276-2. Epub 2019 Aug 16. PMID 31427174
- [Background] Park DE, Higdon MM, Prosperi C, Baggett HC, Brooks WA, Feikin DR, Hammitt LL, Howie SRC, Kotloff KL, Levine OS, Madhi SA, Murdoch DR, O'Brien KL, Scott JAG, Thea DM, Antonio M, Awori JO, Baillie VL, Bunthi C, Kwenda G, Mackenzie GA, Moore DP, Morpeth SC, Mwananyanda L, Paveenkittiporn W, Ziaur Rahman M, Rahman M, Rhodes J, Sow SO, Tapia MD, Deloria Knoll M. Upper Respiratory Tract Co-detection of Human Endemic Coronaviruses and High-density Pneumococcus Associated With Increased Severity Among HIV-Uninfected Children Under 5 Years Old in the PERCH Study. Pediatr Infect Dis J. 2021 Jun 1;40(6):503-512. doi: 10.1097/INF.0000000000003139. PMID 33883479
- [Background] Chiu CY, Miller SA. Clinical metagenomics. Nat Rev Genet. 2019 Jun;20(6):341-355. doi: 10.1038/s41576-019-0113-7. PMID 30918369
- [Background] Li N, Cai Q, Miao Q, Song Z, Fang Y, Hu B. High-Throughput Metagenomics for Identification of Pathogens in the Clinical Settings. Small Methods. 2021 Jan 4;5(1):2000792. doi: 10.1002/smtd.202000792. Epub 2020 Dec 13. PMID 33614906
- [Background] Zhang YZ, Chen YM, Wang W, Qin XC, Holmes EC. Expanding the RNA Virosphere by Unbiased Metagenomics. Annu Rev Virol. 2019 Sep 29;6(1):119-139. doi: 10.1146/annurev-virology-092818-015851. Epub 2019 May 17. PMID 31100994
- [Background] Wu F, Zhao S, Yu B, Chen YM, Wang W, Song ZG, Hu Y, Tao ZW, Tian JH, Pei YY, Yuan ML, Zhang YL, Dai FH, Liu Y, Wang QM, Zheng JJ, Xu L, Holmes EC, Zhang YZ. A new coronavirus associated with human respiratory disease in China. Nature. 2020 Mar;579(7798):265-269. doi: 10.1038/s41586-020-2008-3. Epub 2020 Feb 3. PMID 32015508
- [Background] Boolchandani M, D'Souza AW, Dantas G. Sequencing-based methods and resources to study antimicrobial resistance. Nat Rev Genet. 2019 Jun;20(6):356-370. doi: 10.1038/s41576-019-0108-4. PMID 30886350
- [Background] Suzuki S, Horinouchi T, Furusawa C. Prediction of antibiotic resistance by gene expression profiles. Nat Commun. 2014 Dec 17;5:5792. doi: 10.1038/ncomms6792. PMID 25517437
- [Background] Antimicrobial Resistance Collaborators. Global burden of bacterial antimicrobial resistance in 2019: a systematic analysis. Lancet. 2022 Feb 12;399(10325):629-655. doi: 10.1016/S0140-6736(21)02724-0. Epub 2022 Jan 19. PMID 35065702
- [Background] Howard A, Reza N, Aston S, Woods B, Gerada A, Buchan I, Hope W, Martson AG. Antimicrobial treatment imprecision: an outcome-based model to close the data-to-action loop. Lancet Infect Dis. 2024 Jan;24(1):e47-e58. doi: 10.1016/S1473-3099(23)00367-5. Epub 2023 Aug 31. PMID 37660712
- [Background] Serpa PH, Deng X, Abdelghany M, Crawford E, Malcolm K, Caldera S, Fung M, McGeever A, Kalantar KL, Lyden A, Ghale R, Deiss T, Neff N, Miller SA, Doernberg SB, Chiu CY, DeRisi JL, Calfee CS, Langelier CR. Metagenomic prediction of antimicrobial resistance in critically ill patients with lower respiratory tract infections. Genome Med. 2022 Jul 12;14(1):74. doi: 10.1186/s13073-022-01072-4. PMID 35818068
- [Background] Shi M, Zhao S, Yu B, Wu WC, Hu Y, Tian JH, Yin W, Ni F, Hu HL, Geng S, Tan L, Peng Y, Song ZG, Wang W, Chen YM, Holmes EC, Zhang YZ. Total infectome characterization of respiratory infections in pre-COVID-19 Wuhan, China. PLoS Pathog. 2022 Feb 17;18(2):e1010259. doi: 10.1371/journal.ppat.1010259. eCollection 2022 Feb. PMID 35176118
- [Background] Charalampous T, Alcolea-Medina A, Snell LB, Williams TGS, Batra R, Alder C, Telatin A, Camporota L, Meadows CIS, Wyncoll D, Barrett NA, Hemsley CJ, Bryan L, Newsholme W, Boyd SE, Green A, Mahadeva U, Patel A, Cliff PR, Page AJ, O'Grady J, Edgeworth JD. Evaluating the potential for respiratory metagenomics to improve treatment of secondary infection and detection of nosocomial transmission on expanded COVID-19 intensive care units. Genome Med. 2021 Nov 17;13(1):182. doi: 10.1186/s13073-021-00991-y. PMID 34784976
- [Background] Metlay JP, Waterer GW, Long AC, Anzueto A, Brozek J, Crothers K, Cooley LA, Dean NC, Fine MJ, Flanders SA, Griffin MR, Metersky ML, Musher DM, Restrepo MI, Whitney CG. Diagnosis and Treatment of Adults with Community-acquired Pneumonia. An Official Clinical Practice Guideline of the American Thoracic Society and Infectious Diseases Society of America. Am J Respir Crit Care Med. 2019 Oct 1;200(7):e45-e67. doi: 10.1164/rccm.201908-1581ST. PMID 31573350
- [Background] Harris M, Clark J, Coote N, Fletcher P, Harnden A, McKean M, Thomson A; British Thoracic Society Standards of Care Committee. British Thoracic Society guidelines for the management of community acquired pneumonia in children: update 2011. Thorax. 2011 Oct;66 Suppl 2:ii1-23. doi: 10.1136/thoraxjnl-2011-200598. PMID 21903691
- [Background] Li ZJ, Zhang HY, Ren LL, Lu QB, Ren X, Zhang CH, Wang YF, Lin SH, Zhang XA, Li J, Zhao SW, Yi ZG, Chen X, Yang ZS, Meng L, Wang XH, Liu YL, Wang X, Cui AL, Lai SJ, Jiang T, Yuan Y, Shi LS, Liu MY, Zhu YL, Zhang AR, Zhang ZJ, Yang Y, Ward MP, Feng LZ, Jing HQ, Huang LY, Xu WB, Chen Y, Wu JG, Yuan ZH, Li MF, Wang Y, Wang LP, Fang LQ, Liu W, Hay SI, Gao GF, Yang WZ; Chinese Centers for Disease Control and Prevention (CDC) Etiology of Respiratory Infection Surveillance Study Team. Etiological and epidemiological features of acute respiratory infections in China. Nat Commun. 2021 Aug 18;12(1):5026. doi: 10.1038/s41467-021-25120-6. PMID 34408158
- [Result] Alcock BP, Raphenya AR, Lau TTY, Tsang KK, Bouchard M, Edalatmand A, Huynh W, Nguyen AV, Cheng AA, Liu S, Min SY, Miroshnichenko A, Tran HK, Werfalli RE, Nasir JA, Oloni M, Speicher DJ, Florescu A, Singh B, Faltyn M, Hernandez-Koutoucheva A, Sharma AN, Bordeleau E, Pawlowski AC, Zubyk HL, Dooley D, Griffiths E, Maguire F, Winsor GL, Beiko RG, Brinkman FSL, Hsiao WWL, Domselaar GV, McArthur AG. CARD 2020: antibiotic resistome surveillance with the comprehensive antibiotic resistance database. Nucleic Acids Res. 2020 Jan 8;48(D1):D517-D525. doi: 10.1093/nar/gkz935. PMID 31665441